CLINICAL TRIAL: NCT03832010
Title: Proof of Concept Investigation of the Steroid-reducing Effects of Crisaborole in Children
Brief Title: Steroid-reducing Effects of Crisaborole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00178631
Record Dates: First submitted 2019-01-25; First posted 2019-02-06 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Topical steroid; Crisaborole; Topical calcineurin inhibitor
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — crisaborole; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Crisaborole (Active Comparator): Participants will be instructed to apply emollient, topical steroid, and or crisaborole (blinded) to affected areas with eczema.
  Interventions: Drug: Crisaborole; Drug: Hydrocortisone Ointment; Drug: Triamcinolone ointment; Drug: Aquaphor
- Vehicle (Placebo Comparator): Participants will be instructed to apply emollient, topical steroid, and or vehicle (blinded) to affected areas with eczema.
  Interventions: Drug: Hydrocortisone Ointment; Drug: Triamcinolone ointment; Drug: Aquaphor
- Control (Sham Comparator): Participants will be instructed to apply emollient, topical steroid, and or emollient (blinded) to affected areas with eczema.
  Interventions: Drug: Hydrocortisone Ointment; Drug: Triamcinolone ointment; Drug: Aquaphor

INTERVENTIONS:
Drug: Crisaborole — Participants will be instructed to apply crisaborole to affected areas with eczema.
  Other Names: Eucrisa
  Arms: Crisaborole
Drug: Hydrocortisone Ointment — Participants will be instructed to apply hydrocortisone to affected areas with eczema on face, armpits or groin.
Drug: Triamcinolone ointment — Participants will be instructed to apply triamcinolone to affected areas on the body excluding face, armpits or groin.
Drug: Aquaphor — Participants will be instructed to moisturize all over the body with Aquaphor.

SUMMARY:
Atopic dermatitis, or eczema, is a chronic skin condition affecting many children. Crisaborole is a non-steroid topical medication which is FDA approved for children aged 2 and older for eczema. This research study seeks to investigate whether crisaborole reduces topical steroid use in children with atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic skin disease and a common affliction among children. Twice daily topical corticosteroid (TCS) use over several weeks is recommended for active inflammatory disease. Side effects of TCS range from cutaneous atrophy to hypothalamic-pituitary-adrenal axis suppression. Steroid phobia and misunderstanding often lead to poor compliance and inadequate disease control. Topical calcineurin inhibitors (TCIs) are currently recommended as steroid-reducing agents, especially on sensitive areas such as the face and skin folds. However, TCis are associated with burning reactions and come with black box warnings.

Crisaborole (Eucrisa), the newest topical prescription option for AD, is a phosphodiesterase-4 inhibitor with demonstrated efficacy in patients aged 2 and older with mild to moderate AD. Given the good tolerability and favorable safety profile, crisaborole makes for an alternative topical option to its predecessors. However, corresponding data are lacking. It would be of great interest to patients, patients' families and providers if crisaborole can be shown to reduce the amount of TCS necessary for control of AD. The investigators therefore propose a proof-of-concept study to investigate whether crisaborole can serve as an effective steroid-reducing agent.

ELIGIBILITY:
Inclusion criteria:

* Children aged 2 or older (<18).
* Diagnosed with atopic dermatitis.
* At baseline, AD is mild to moderate (score of 2 [mild] to 3 [moderate]) on the Investigator's Global Assessment scale (IGA; scores range 0-4, higher indicates greater severity).

Exclusion criteria:

* Known allergy to a constituent of the studied products (crisaborole, vehicle, Aquaphor, topical steroids [hydrocortisone 2.5% ointment and triamcinolone acetonide 0.1% ointment]).
* At baseline, AD is severe (score of 4 [severe] on the IGA scale).
* Medical problems which interfere with completion of protocols in this study.
* Pregnant or lactating females. (Females who have experienced menarche will be required to take a urine pregnancy test.)
* Participant is enrolled in another research study.
* Participant or participant's guardian(s) are unable to follow instructions as required in this study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Grossberg, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paller AS, Tom WL, Lebwohl MG, Blumenthal RL, Boguniewicz M, Call RS, Eichenfield LF, Forsha DW, Rees WC, Simpson EL, Spellman MC, Stein Gold LF, Zaenglein AL, Hughes MH, Zane LT, Hebert AA. Efficacy and safety of crisaborole ointment, a novel, nonsteroidal phosphodiesterase 4 (PDE4) inhibitor for the topical treatment of atopic dermatitis (AD) in children and adults. J Am Acad Dermatol. 2016 Sep;75(3):494-503.e6. doi: 10.1016/j.jaad.2016.05.046. Epub 2016 Jul 11. PMID 27417017
- [Background] Eichenfield LF, Tom WL, Berger TG, Krol A, Paller AS, Schwarzenberger K, Bergman JN, Chamlin SL, Cohen DE, Cooper KD, Cordoro KM, Davis DM, Feldman SR, Hanifin JM, Margolis DJ, Silverman RA, Simpson EL, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Sidbury R. Guidelines of care for the management of atopic dermatitis: section 2. Management and treatment of atopic dermatitis with topical therapies. J Am Acad Dermatol. 2014 Jul;71(1):116-32. doi: 10.1016/j.jaad.2014.03.023. Epub 2014 May 9. PMID 24813302

RESULTS

PARTICIPANT FLOW:
Groups:
- Crisaborole: Crisaborole is chosen because it is the newest non-steroid FDA-approved prescription topical medication for treatment of mild to moderate AD in children 2 years of age and older. The FDA-approved dosage is application of a thin layer twice daily to affected areas.
  Hydrocortisone and triamcinolone are chosen because these are commonly prescribed topical steroids for treatment of mild to moderate AD in children 2 years of age and older. Hydrocortisone is a low-potency topical steroid, and triamcinolone is a mid-potency topical steroid. The FDA-approved dosage for hydrocortisone and triamcinolone is application of a thin layer twice daily to affected areas.
  Crisaborole: Participants will be instructed to apply crisaborole to affected areas with eczema.
  In the crisaborole group, the parents will be provided with crisaborole (with unidentifiable packaging) with refills as needed. As for twice daily topical corticosteroid (TCS), triamcinolone acetonide 0.1% ointment and hydrocortisone 2.5% ointment will be provided, with refills as needed. Aquaphor is to be applied for maintenance. Crisaborole will be used as the first-line agent for AD lesions. TCS will be used as the second-line agent for AD lesions.
- Vehicle: Crisaborole vehicle is chosen because this contains only the inactive ingredients found in crisaborole, to serve as placebo.
  Hydrocortisone and triamcinolone are chosen because these are commonly prescribed topical steroids for treatment of mild to moderate AD in children 2 years of age and older. Hydrocortisone is a low-potency topical steroid, and triamcinolone is a mid-potency topical steroid. The FDA-approved dosage for hydrocortisone and triamcinolone is application of a thin layer twice daily to affected areas.
  In the vehicle group, parents will be provided vehicle (non-medicated ointment) with unidentifiable packaging, with refills as needed. They will also have triamcinolone acetonide 0.1% ointment and hydrocortisone 2.5% ointment provided, with refills as needed. They will be provided identical instructions to the crisaborole group with regard to usage of the vehicle and TCS.
- Control: Aquaphor is chosen because this is a skin moisturizer which is routinely used by patients with AD.
  Hydrocortisone and triamcinolone are chosen because these are commonly prescribed topical steroids for treatment of mild to moderate AD in children 2 years of age and older. Hydrocortisone is a low-potency topical steroid, and triamcinolone is a mid-potency topical steroid. The FDA-approved dosage for hydrocortisone and triamcinolone is application of a thin layer twice daily to affected areas.
  In the control group, parent(s) will be provided control (Aquaphor) in unidentifiable packaging, with refills as needed. They will also be provided triamcinolone acetonide 0.1% ointment and hydrocortisone 2.5% ointment, with refills as needed. They will be given identical instructions to the crisaborole and vehicle groups with regard to usage of TCS.
Period: Overall Study
Arm/Group | Crisaborole | Vehicle | Control
Started | 8 | 7 | 9
Completed | 4 | 5 | 8
Not Completed | 4 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crisaborole | Vehicle | Control | Total
Number analyzed (Participants) | 8 | 7 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.88 (5.17) | 7.86 (3.93) | 6.56 (3.81) | 7.375 (4.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 15
  Male | 3 | 3 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 3 | 6
  White | 7 | 2 | 5 | 14
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Steroid Usage Quantity
Description: Steroid usage measured in medication weight (grams)
Time Frame: Day 30
Population: 3 withdrew, 7 lost to followup
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 4 | 5 | 5
grams | 7.27 (10.00) | 10.78 (20.77) | 8.22 (10.39)

2. Primary Outcome: Steroid Usage Quantity
Description: Steroid usage measured in medication weight (grams)
Time Frame: Day 90
Population: 3 withdrew, 9 lost to followup
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 2 | 4 | 6
grams | 37.82 (27.49) | 16.15 (18.79) | 5.43 (11.13)

3. Primary Outcome: Steroid Usage Frequency
Description: Steroid usage measured in diary entries. Weekly average frequency of steroid use is reported.
Time Frame: Day 30
Measure: Mean (Standard Deviation); unit: steroids used per week
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 5 | 5 | 8
steroids used per week | 1.81 (1.41) | 1.27 (1.21) | 1.85 (1.09)

4. Primary Outcome: Steroid Usage Frequency
Description: Steroid usage measured in diary entries. Weekly average frequency of steroid use is reported.
Time Frame: Day 90
Population: Participants lost to follow-up in recording diaries, data not collected.
Measure: Mean (Standard Deviation); unit: steroids used per week
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 3 | 5 | 8
steroids used per week | 2.74 (3.62) | 1.71 (1.80) | 1.38 (1.11)

5. Secondary Outcome: Eczema Severity as Assessed by SCORing Atopic Dermatitis (SCORAD) Score
Description: Clinical assessment using SCORAD score: minimum score = 0, maximum score = 103. Highest score corresponds with highest severity of eczema. Lowest score corresponds with lowest severity of eczema.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 8 | 7 | 9
score on a scale | 29.15 (10.79) | 28.75 (9.68) | 29.04 (14.43)

6. Secondary Outcome: Eczema Severity Assessed by SCORAD Score
Description: Clinical assessment using SCORAD score: minimum score = 0, maximum score = 103. Higher score corresponds with increased severity of eczema. Lowest score corresponds with lowest severity of eczema.
Time Frame: Day 30
Population: There were some lost-to-follow up after Day 0.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 5 | 5 | 7
score on a scale | 26.88 (9.64) | 25.40 (17.49) | 22.66 (8.21)

7. Secondary Outcome: Eczema Severity Assessed by SCORAD Score
Description: as for outcome 6
Time Frame: Day 90
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 4 | 5 | 8
score on a scale | 25.78 (7.90) | 17.20 (8.74) | 18.99 (10.66)

8. Secondary Outcome: Quality of Life for Participant as Assessed by Children's Dermatology Life Quality Index
Description: Children's Dermatology Life Quality Index (ages 15 or younger). The minimum score is 0, maximum score is 30. The highest score corresponds with most severe impairment of quality of life. The lowest score corresponds with lowest impairment of quality of life.
Time Frame: Day 0
Population: Some participants were lost to follow-up, data not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 6 | 6 | 9
score on a scale | 10.67 (5.65) | 4.67 (4.50) | 8.89 (5.99)

9. Secondary Outcome: Quality of Life for Participant as Assessed by Children's Dermatology Life Quality Index
Description: as for outcome 8
Time Frame: Day 30
Population: Some participants were lost to follow-up, data not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 4 | 6 | 8
score on a scale | 5 (2.83) | 3.17 (5.38) | 4.63 (4.93)

10. Secondary Outcome: Quality of Life for Participant as Assessed by Children's Dermatology Life Quality Index
Description: as for outcome 8
Time Frame: Day 90
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 4 | 5 | 8
score on a scale | 5.75 (2.5) | 2 (1.58) | 3.625 (4.37)

11. Secondary Outcome: Quality of Life for Family as Assessed by Dermatitis Family Impact Questionnaire
Description: Dermatitis Family Impact Questionnaire. Minimum score is 0, maximum score is 30. The highest score corresponds with most severe impairment of quality of life. The lowest score corresponds with lowest impairment of quality of life.
Time Frame: Day 0
Population: Some participants were lost to follow-up, data not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 6 | 6 | 9
score on a scale | 11.17 (5.12) | 6.67 (6.83) | 7.89 (6.72)

12. Secondary Outcome: Quality of Life for Family as Assessed by Dermatitis Family Impact Questionnaire
Description: as for outcome 11
Time Frame: Day 30
Population: Some participants were lost to follow-up, data not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 4 | 6 | 8
score on a scale | 7 (4.97) | 5.5 (9.18) | 3.125 (2.75)

13. Secondary Outcome: Quality of Life for Family as Assessed by Dermatitis Family Impact Questionnaire
Description: as for outcome 11
Time Frame: Day 90
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 4 | 5 | 8
score on a scale | 10.25 (11.53) | 2.6 (3.71) | 3.125 (3.72)

14. Secondary Outcome: Severity of Itching as Assessed by Pruritus Score
Description: Pruritus score determined using Numerical Rating Scale. Minimum score is 0. Maximum score is 10. Lowest score means no itching. Highest score corresponds to the most severe itching imaginable by patient.
Time Frame: Day 0
Population: Some participants were lost to follow-up, data not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 8 | 7 | 8
score on a scale | 5.25 (2.71) | 5.71 (3.35) | 5.25 (2.60)

15. Secondary Outcome: Severity of Itching as Assessed by Pruritus Score
Description: as for outcome 14
Time Frame: Day 30
Population: Some participants were lost to follow-up, data not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 5 | 6 | 8
score on a scale | 5.2 (1.30) | 4.17 (2.93) | 3.125 (1.89)

16. Secondary Outcome: Severity of Itching as Assessed by Pruritus Score
Description: as for outcome 14
Time Frame: Day 90
Population: Some participants were lost to follow-up, data not collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Vehicle | Control
Number analyzed (Participants) | 3 | 5 | 8
score on a scale | 4 (1.73) | 2.8 (2.17) | 2.125 (2.42)

ADVERSE EVENTS:
Time Frame: Up to 104 days
Arm/Group | Crisaborole | Vehicle | Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 1/8 | 0/7 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crisaborole (N=8) | Vehicle (N=7) | Control (N=9)
burning sensation after the first application of the assigned study medication. (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT03832010/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT03832010/ICF_001.pdf